CLINICAL TRIAL: NCT01321944
Title: A POPULATION-BASED DIRECT-TO-SMOKER OUTREACH OFFERING TOBACCO TREATMENT IN A HEALTH CARE SETTING: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Direct to Smoker Outreach in a Health Care Setting
Acronym: DTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Partners HealthCare, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Nancy Rigotti, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P001137
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual clinical care (No Intervention): Usual clinical care provided by health care system
- DTS intervention (Experimental): Intervention group participants will be sent 3 letters at monthly intervals signed by the participant's PCP that encourages the smoker to quit, and offers a free telephone consultation by Partners' Tobacco Treatment Coordinator (TTC), free nicotine patches, and referral to additional treatment resources including the state's free telephone quitline.
  Interventions: Other: Direct to Smoker Outreach Program

INTERVENTIONS:
Other: Direct to Smoker Outreach Program — Intervention group participants will be sent 3 letters at monthly intervals signed by the participant's PCP, encouraging the smoker to quit, and offering a free telephone consultation by Partners' Tobacco Treatment Coordinator (TTC). Participants can respond to the treatment offer by calling or emailing the TTC, who will provide a 15-minute consultation following the "5A" strategy recommended by the US Public Health Service's clinical guideline and help smokers access treatment by (1) offering a free 4-week supply of 21mg nicotine patches sent by secure mailing to their home (refillable once for a total of 8 weeks), (2) helping smokers obtain prescriptions from their PCP for other FDA-approved smoking cessation medication, (3) using a fax-referral system to facilitate connection to free multi-session counseling from the Massachusetts Smokers Quitline, and (4) referring to local in-person counseling programs.
  Other Names: Nicotine transdermal patch
  Arms: DTS intervention

SUMMARY:
Tobacco use is the leading preventable cause of death in the United States. Effective treatment for tobacco dependence exists and includes counseling and pharmacotherapy with nicotine replacement, bupropion, or varenicline. The health care system is a key channel for delivering this treatment to smokers. Brief clinical interventions delivered at office visits increase smoking cessation rates, are among the most cost-effective of medical interventions, and are recommended by U.S. Public Health Service. However, physicians and other clinicians often fail to provide them. Clinicians' rates of providing tobacco treatment in ambulatory care can be improved, but even when successful, clinicians can only reach smokers who make an office visit.

A health care system might improve its delivery of tobacco treatment by supplementing visit-based efforts with a population-based strategy, using methods proven effective in public health settings. A population of smokers could be identified from electronic health records and offered treatment proactively in a way that maximizes convenience and minimizes barriers such the cost of pharmacotherapy. This study tests the effectiveness of a population-based Direct-to-Smoker (DTS) outreach program provided to smokers in one community health center in Revere, MA, that is part of an integrated health care system. It uses the system's population management tools to identify smokers and proactively offers them evidence-based tobacco treatment that is free and does require making an office visit. A randomized controlled trial will compare the effectiveness of the DTS program to usual primary care. The hypothesis is that adding the DTS program to usual primary care will increase the proportion of smokers who use tobacco dependence treatment and thereby stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>= 18 years)
* made an office visit to a primary care physician (PCP) at Revere Health Center in the year prior to May 2009
* has a telephone
* listed as a smoker in the past 5 years in the electronic health record

Exclusion Criteria:

* severe psychiatric or neurologic diagnosis (e.g., psychosis, dementia) on problem list of electronic health record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
proportion of participants who reported using any tobacco dependence treatment during the 3-month study period | 3 months
  Tobacco dependence treatment is defined as (1) any smoking cessation counseling contact (with the Tobacco Treatment Coordinator, the Massachusetts Smokers Quitline, or in-person counseling) or (2) any FDA-approved smoking cessation pharmacotherapy (nicotine patch, gum, lozenge, inhaler, or nasal spray; bupropion; or varenicline).

SECONDARY OUTCOMES:
7-day point prevalence abstinence from tobacco products | 3 month follow-up
  tobacco abstinence, defined as self-reported 7-day point prevalence abstinence at 3-month follow-up
30-day point prevalence abstinence from tobacco products | 3 month follow-up
  Tobacco abstinence, defined as self-reported 30-day point prevalence abstinence at 3-month follow-up
Use of nicotine replacement therapy | Past 3 months
  Use of nicotine patch, gum, lozenge, inhaler, or nasal spray in the past 3 months.
Use of any tobacco cessation medication | Past 3 months
  Use of any nicotine replacement product, varenicline, or bupropion in the past 3 months in order to quit smoking
Use of smoking cessation counseling | Past 3 months
  Use of telephone or in-person smoking cessation counseling in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Revere Health Center, Revere, Massachusetts, United States

REFERENCES:
- [Derived] Rigotti NA, Bitton A, Kelley JK, Hoeppner BB, Levy DE, Mort E. Offering population-based tobacco treatment in a healthcare setting: a randomized controlled trial. Am J Prev Med. 2011 Nov;41(5):498-503. doi: 10.1016/j.amepre.2011.07.022. PMID 22011421